CLINICAL TRIAL: NCT04529551
Title: CSD1601: A Crossover Study to Evaluate the Exposure to Tar and Nicotine From Two Cigarette Products That Contain a Menthol Capsule in the Filter
Brief Title: CSD1601: A Study to Evaluate the Exposure to Tar and Nicotine From Two Cigarette Products That Contain a Menthol Capsule in the Filter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAI Services Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CSD1601
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Smoking; Tobacco Smoking; Tobacco Use
MeSH Terms: conditions — Smoking; Tobacco Smoking; Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1601A, 1601B product use order (Experimental): Subjects will use 1601A for 1 week and then 1601B for 1 week.
  Interventions: Other: 1601A; Other: 1601B
- 1601B, 1601A product use order (Experimental): Subjects will use 1601B for 1 week and then 1601A for 1 week.
  Interventions: Other: 1601A; Other: 1601B

INTERVENTIONS:
Other: 1601A — A filtered, king size cigarette with a menthol capsule in the filter.
Other: 1601B — A filtered, king size cigarette with a menthol capsule in the filter.

SUMMARY:
This study will evaluate exposure to tar and nicotine from two cigarette products that contain a menthol capsule in the filter, and provide a basis for comparing mouth-level exposure when smokers smoke the two cigarette products.

DETAILED DESCRIPTION:
Subjects will be randomly assigned to the order in which they will smoke two study cigarette products (including one comparator product and one test product). Subjects will smoke each study product exclusively for approximately one week prior to a test visit, with a different product smoked each week over a two-week period. Cigarette butts will be collected the day prior to each test visit for determination of Yield-in-Use (YIU) tar and nicotine levels. Blood samples will be collected at each test visit for determination of blood cotinine levels. Subjects will provide responses to questions during each test visit to assess their cigarette smoking and cigarette butt collection behavior during the preceding day.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and willing to sign an Informed Consent Form (ICF) written in English;
2. Generally healthy males and females, 21 years of age or older, at Screening- Enrollment Visit;
3. Self-reports smoking at least seven cigarettes per day and inhaling the smoke;
4. Usual brand of cigarette is one of the brand styles specified;
5. Smoked usual brand for ≥ 3 months;
6. Subject does not intend to delay a decision to quit smoking to participate in the study.
7. Agrees to exclusively smoke the study cigarettes and not smoke or use any other tobacco or nicotine-containing products during the course of the study.
8. Able to read and comprehend English.
9. Able to safely perform the required study procedures, as determined by the Investigator.

Exclusion Criteria:

1. Self-reported history of heart disease, kidney disease, asthma or any other lung disease, diabetes, liver disease, hypertension, or hypercholesterolemia.
2. At risk for heart disease, i.e., obesity (body mass index [BMI] ≥ 40 kg/m2), as determined by the Investigator;
3. Females ≥ 35 years of age currently using systemic, estrogen-containing contraception, or hormone replacement therapy;
4. Postponing a decision to quit smoking (defined as planning a quit attempt within 30 days of the Screening-Enrollment Visit) to participate in this study;
5. Use of any medication or substance that aids in smoking cessation, including but not limited to any nicotine-replacement therapy (NRT) (e.g., nicotine gum, lozenge, patch), varenicline (Chantix®), bupropion (Wellbutrin®, Zyban®), or lobelia extract within 30 days prior to the Screening-Enrollment Visit;
6. Females who test positive for pregnancy, are pregnant or breastfeeding, or plan to become pregnant during the course of the study;
7. Determined by the Investigator to be inappropriate for the study;

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-04-08 (Actual); Primary Completion 2016-05-02 (Actual); Study Completion 2016-05-02 (Actual)

PRIMARY OUTCOMES:
Yield-in-use tar per cigarette | 2 weeks
  To compare the per cigarette YIU tar per cigarette from smoking product 1601A with those from smoking product 1601B.
Yield-in-use nicotine per cigarette | 2 weeks
  To compare the per cigarette YIU nicotine per cigarette from smoking product 1601A with those from smoking product 1601B.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Austin, MD, Principal Investigator — High Point Clinical Trials Center
Locations (1):
- High Point Clinical Trials Center, High Point, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No